CLINICAL TRIAL: NCT04739345
Title: Effect of Pentoxifylline on Immune-inflammation Index for Predicting Prognosis of Coronavirus Disease 2019 (COVID- 19) Infection
Brief Title: Effect of Pentoxifylline on Prognosis of Coronavirus Disease 2019 (COVID- 19) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer at Faculty of Pharmacy, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-Pentoxifylline
Record Dates: First submitted 2021-02-03; First posted 2021-02-04 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Corona Virus Infection; Cytokine Storm
Keywords: COVID-19; Cytokine Storm; Interleukin-6
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Cytokine Release Syndrome | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Non-severe patients should meet all following conditions: (1) Epidemiology history, (2) Fever or other respiratory symptoms, (3) Typical CT image abnormities of viral pneumonia, and (4) Positive result of RT-PCR for SARS-CoV-2 RNA.
  Interventions: Drug: Pentoxifylline
- Group 2 (Placebo Comparator): Severe patients should meet at least one of the following conditions: (1) Shortness of breath, RR ≥ 30 times/min, (2) Oxygen saturation (Resting state) ≤ 93%, (3) PaO2/FiO2 ≤ 300 mmHg.
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — 400 mg of pentoxifylline orally TID with the standard COVID-19 protocol of the Egyptian Ministry of Health

SUMMARY:
Coronavirus disease 2019 (COVID-19) remains a threatening pandemic, due to its rapid transmission, uncertain risk factors for progression that lead to its lethality and yet unsatisfactory antiviral therapy or prophylaxis. The respiratory system remains the most frequently affected by the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2), with patients either presenting mild illness as well as more severe complications such as acute respiratory distress syndrome (ARDS) that necessitates admission in Intensive Care Units (ICU). Unfortunately, the remaining patients progress to a second phase-called the inflammatory stage-featuring ARDS, thromboembolic events, and myocardial acute injury. These clinical exacerbation latter predicts poor prognosis associated with an exacerbation of the immune system cascade; a phenomenon known as "cytokine storm". In the context of COVID-19, the hyper inflammation diagnostic criteria are partly defined. Early studies of patients with COVID-19 established independent associations between biomarkers of inflammation, such as C-reactive protein, interleukin [IL]-6, ferritin and D-dimer, and severe disease states that require respiratory support or result in death.

The aim of this study was to identify practical blood immune- inflammatory biomarker / ratio that could be used alternatively to IL-6 for predicting severity of coronavirus disease 2019 (COVID- 19) in clinical practice.

Another aim is to unveil the association of the pro-inflammatory profile as categorized by the IL-6 levels in patients infected by SARS-COV-2, with disease severity and outcomes of COVID -19.

DETAILED DESCRIPTION:
Recent research confirmed that levels of IL-6 seem are associated with COVID-19 induced inflammatory response, respiratory failure, needing for mechanical ventilation and/or intubation and mortality. The importance of identifying Il-6 as a biomarker lies in the potential use of antibody against IL-6 such as tocilizumab, which is currently used in the treatment protocol of covid-19. The authors shared an encouraging experience of utilizing tocilizumab medication, particularly in patients at risk of developing chemokine storm secondary to COVID-19. IL-6, a chemokine, is an important biomarker of inflammation and has been shown in studies as an important predictor of severe COVID-19. IL-6 is responsible for elevation of acute phase reactants, such as C-reactive protein, serum amyloid A, fibrinogen, and hepcidin, and inhibition of albumin synthesis. The dysregulated production of IL-6 has been attributed to autoimmunity and chronic inflammation.

We performed a systematic review and meta analysis to compare IL-6 in severe and non severe patients. In clinical practice, it remains crucial to develop a scoring system that includes IL-6 to assist clinicians in early recognition of patients at risk for developing severe disease.

Circulating biomarker like neutrophil (NEU)-to-lymphocyte (LYM) ratio (NLR) as well as other ratios are used to represent inflammation and the immune status and are considered a potential predictor for the prognosis of COVID-19 patients. Interestingly clinical scores like the CALL score (C = comorbidity, A= age, L = lymphocyte count, L = lactate dehydrogenase (LDH)) have been used for predicting progression towards clinical worsening.

Adding IL-6 levels to the CALL score proved to improve its predictive power and make treatment more appropriate, especially in patients for whom decision whether to treat or not with IL-6 inhibitors such as tocilizumab is required. It should be recognized that the CALL-IL-6 score could be difficult to reproduce in low- and medium-income countries due to costs of IL-6 dosage.

Aim of the Study

1. Identify new blood immune inflammatory biomarker / ratio that could be used alternatively to IL-6 for predicting severity of coronavirus disease 2019 (COVID- 19) in clinical practice.
2. Evaluate the influence of the pro-inflammatory profile on clinical outcomes and therapeutic efficacy as categorized by the IL-6 levels in patients infected by SARS-COV-2.
3. Assess potential associations with other blood inflammatory biomarker and the impact of the inflammatory status on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years.
2. COVID-19 hospitalized patients with pneumonia proved by chest X-ray or CT scan.
3. Confirmed infection with COVID-19 virus using RT-PCR or strongly suspected to be infected with pending confirmation studies.
4. Have acute respiratory distress syndrome (ARDS).
5. Having either peripheral capillary oxygen saturation (SpO2) ≤ 94% ambient air, or a partial oxygen pressure (PaO2) to fraction of inspired oxygen (FiO2) ratio ≤ 300 mmHg.

Exclusion Criteria:

1. Age greater than 85 years-old
2. Creatinine clearance (CrCl) < 10ml/min.
3. Severe circulatory shock with a dose of norepinephrine higher than 1.0 μg/kg/min.
4. Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in patients' clinical status | Two weeks
  Change in clinical status will be assessed daily using six category ordinal scale. The categories were defined as follows: 1) patient discharged, 2) hospitalization not requiring supplemental oxygen, 3) hospitalization requiring supplemental low-flow oxygen, 4) hospitalization requiring high-flow supplemental oxygen, 5) hospitalization requiring invasive mechanical ventilation, 6) death.
Time to increase in oxygenation | 48 hours
  Time to increase in SpO2/FiO2 of 50 or greater compared to the baseline SpO2/FiO2
Duration of hospitalization | Two weeks
  Length of hospital stay
In hospital mortality | Two weeks
  Death occurrence during hospitalization

SECONDARY OUTCOMES:
Incidence of non-invasive mechanical ventilation | Two weeks
  Need for non-invasive mechanical ventilation
Duration of non-invasive mechanical ventilation | Two weeks
  Time required on non-invasive mechanical ventilation
Incidence of invasive mechanical ventilation | Two weeks
  Need for invasive mechanical ventilation
Duration of invasive mechanical ventilation | Two weeks
  Time required on invasive mechanical ventilation
Occurrence of secondary infection | Two weeks
  Occurrence of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Neven Sarhan, PhD, Principal Investigator — Misr International University
Locations (1):
- Teachers Hospital, Cairo, Please Select, Egypt

IPD SHARING:
Plan to Share IPD: No